CLINICAL TRIAL: NCT05530278
Title: Assessment of Multiple-Dose Pharmacokinetics and Safety of the Co-administration of Galicaftor, Navocaftor and ABBV-576 and Potential of ABBV-576 for CYP3A Induction in Healthy Volunteers
Brief Title: A Study to Assess the Pharmacokinetics and Safety of Co-administered Oral Galicaftor, Navocaftor, and ABBV-576 in Healthy Adults for the Treatment of Cystic Fibrosis
Acronym: ABBV-576 DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20-974
Record Dates: First submitted 2022-09-05; First posted 2022-09-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
Keywords: Galicaftor; Navocaftor; ABBV-576; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- ABBV-576 with Galicaftor + Navocaftor (Experimental): Participants will receive ABBV-576 for 14 consecutive days, with navocaftor + galicaftor for the latter 7 consecutive days.
  Interventions: Drug: Galicaftor; Drug: ABBV-576; Drug: Navocaftor
- Navocaftor + Galicaftor with ABBV 576 (Experimental): Participants will receive Navocaftor + galicaftor for 14 consecutive days, with ABBV 576 for the latter 7 consecutive days.
  Interventions: Drug: Galicaftor; Drug: ABBV-576; Drug: Navocaftor
- Optional: Navocaftor with ABBV 576 (Experimental): Participants will receive Navocaftor for 14 consecutive days with ABBV 576 for the latter 7 consecutive days.
  Interventions: Drug: ABBV-576; Drug: Navocaftor
- Optional: Galicaftor with ABBV 576 (Experimental): Participants will receive Galicaftor for 14 consecutive days, with ABBV 576 for the latter 7 consecutive days.
  Interventions: Drug: Galicaftor; Drug: ABBV-576
- Optional: Midazolam with ABBV-576 + Navocaftor (Experimental): Participants will receive Midazolam alone and in combination with multiple doses of ABBV-576 + navocaftor.
  Interventions: Drug: ABBV-576; Drug: Navocaftor; Drug: Midazolam

INTERVENTIONS:
Drug: Galicaftor — Oral
  Arms: ABBV-576 with Galicaftor + Navocaftor; Navocaftor + Galicaftor with ABBV 576; Optional: Galicaftor with ABBV 576
Drug: ABBV-576 — Oral
Drug: Navocaftor — Oral
  Arms: ABBV-576 with Galicaftor + Navocaftor; Navocaftor + Galicaftor with ABBV 576; Optional: Midazolam with ABBV-576 + Navocaftor; Optional: Navocaftor with ABBV 576
Drug: Midazolam — Oral
  Arms: Optional: Midazolam with ABBV-576 + Navocaftor

SUMMARY:
Cystic Fibrosis (CF) is a rare, life-threatening, genetic disease that affects the lungs and digestive system, significantly impairing the quality of life, with those affected having a median age of death at 40. The main objectives of this study are to assess the safety and pharmacokinetics of the combination therapy of galicaftor/navocaftor/ABBV-576.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is ≥ 18.0 to ≤ 29.9 kg/m2 after rounding to the tenths decimal.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication or food.
* History of any clinically significant condition listed in the protocol.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to Day 52
  Cmax will be assessed.
Time to maximum observed plasma concentration (Tmax) | Up to Day 52
  Tmax will be assessed.
Apparent terminal phase elimination rate constant (BETA or β) | Up to Day 52
  Apparent terminal phase elimination rate constant (BETA or β) will be assessed.
Mean terminal phase elimination half-life (t1/2) | Up to Day 52
  T1/2 will be assessed.
Area under the plasma curve (AUC) | Up to Day 52
  AUC will be assessed.
Number of Participants With Adverse Events (AEs) | Up to Day 82
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - Anaheim Clinical Trials LLC /ID# 248824, Anaheim, California
  - Clinical Pharmacology of Miami /ID# 248823, Miami, Florida
  - PPD Clinical Research Unit -Las Vegas /ID# 248853, Las Vegas, Nevada
  - PPD Clinical Research Unit - Austin /ID# 248854, Austin, Texas

IPD SHARING:
Plan to Share IPD: No